CLINICAL TRIAL: NCT05870137
Title: A Pilot Randomised Cross-over Trial of HoloLens2™️ for the Delivery of Distributed Medical Care During COVID-19 in a Simulated Environment.
Brief Title: Assessing Mixed Reality for Emergency Medical Care Delivery in a Simulated Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 21SM6714
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Emergency Medicine
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised cross-over trial
Who Masked: Outcomes Assessor
Masking Description: To ensure masking in this clinical trial, the intervention sequence was randomized for each participant, and the assessors were kept blinded to the sequence. The assessors were not informed about which intervention was provided to each participant or which arm of the study each participant completed first.
  The trial achieved masking by randomly allocating participants to either the control or intervention groups and further by anonymizing the data after capturing the sequence, prior to releasing it to the outcome assessors. This approach ensured that the assessors were not biased in their assessments and were unaware of which intervention was provided to each participant. By blinding the assessors, the study was able to reduce potential sources of bias and increase the validity and reliability of the results. Overall, the masking approach used in this trial was designed to minimize the risk of bias and ensure that the results were as objective and accurate as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Standard care was delivered by the participants with access to didactic instruction and telephonic support. Participants had access to all resources through standard ward base computer systems. Access to senior support through telephone call using a bleep/on call system standard to practice within the institution.
  Interventions: Other: Standard care
- Mixed reality - HoloLens2TM Supported care (Experimental): HL2 supported care made all of these resources available through interaction with the HL2 device. Participants had access to all resources through the Mixed reality device (HoloLens2). Access to senior support through using the HL2 device.
  Interventions: Device: HoloLens2TM

INTERVENTIONS:
Device: HoloLens2TM — Participants assigned to Mixed Reality-supported care used the HoloLens2 device, which provided support using technology that was permitted by the device. This support included remote assistance and holographic versions of patient-specific investigation results, such as radiological findings, biochemistry, and guidelines for completing the procedure (insertion of chest drain).
  Arms: Mixed reality - HoloLens2TM Supported care
Other: Standard care — The standard care for the intervention involved participants performing the invasive technical procedure to treat a tension pneumothorax using their standard clinical skills and knowledge, without the aid of the HoloLens2 device. The participants in the standard care group did not receive any additional support or guidance beyond what is typically available in a clinical setting. The goal of the study was to compare the effectiveness of the standard care approach with the use of Mixed Reality-supported care using the HoloLens2 device.
  Arms: Standard care

SUMMARY:
This study assessed the feasibility and effectiveness of using Mixed Reality (MR) through the use of HoloLens2TM technology to enhance emergency clinical care delivery in a simulated environment. This was achieved by inviting 22 resident grade doctors to complete two scenarios. Each scenario was supported either by standard care methods or Mixed reality. The participants were randomised to at the start of the scenarios to determine which support they would receive first. The main outcome was to see if there was difference in error rates. This was assessed using the ICECAP multidimensional error capture tool. Secondary outcomes included teamwork, scenario completion, stress/cognitive load, and Mixed reality device user acceptability.

ELIGIBILITY:
Inclusion Criteria:

* All participants must provide consent to participate in the study
* Participants must receive a standardised HL2 headset and operational tutorial
* Participants must complete a qualitative questionnaire to determine their clinical experience and exposure to the technology prior to commencement of the study
* Participants must pass a competency test to ensure standardised basic technical competency and mitigate device related first-use learning effects

Exclusion Criteria:

* Not currently working in emergency medicine/trauma setting
* No prior course completion (Advance trauma and Basic Life support)

Prior to the commencement of the study, all eligible participants were required to provide their consent to participate. Participants were then provided with a standardized HL2 headset and operational tutorial, and completed a qualitative questionnaire to assess their clinical experience and exposure to the technology. The tutorial, which was guided by the research team, included a practical induction providing fundamentals of use, how to make and receive calls, and how to use the clinical data assets provided. Participants were also required to pass a competency test to ensure standardized basic technical competency and mitigate device-related first-use learning effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Error Rate | Through study completion, an average of 8 minutes per scenario
  The primary outcome measure for this study was the error rate, which was assessed using the ICECAP tool (Imperial College Error CAPture). This is a validated, multidimensional tool that assesses errors across several domains, including equipment, communication, technical aspects, patient-related factors, procedure-independent pressures, and a category for capturing any other errors that are not specified. Using the ICECAP tool provides a comprehensive assessment of errors and allows for identifying areas of improvement across multiple domains. Each time an error is observed the participant is attributed 1 score per error within the respective category. The total number of errors is accumulated throughout completion of the scenario. The error is reported as a sum of the total errors observed, as well as per category to determine if there is any specific areas that error rate is impacted.

SECONDARY OUTCOMES:
Scenario completion success | Through study completion, an average of 8 minutes per scenario
  The secondary outcome measure was the successful completion of the clinical scenario. This was determined by the simulation team assessing whether the participant was able to successfully insert the chest drain and complete a life-saving intervention in the simulated environment. If the participant was unable to appropriately insert the chest drain, this was considered an adverse outcome for the simulated patient, and thus the scenario was deemed unsuccessful.
Scenario completion duration | Through study completion, an average of 8 minutes per scenario
  The secondary outcome measure was the time taken to complete the clinical scenario. This was recorded by the simulation team from the initiation of the scenario to the successful completion, which involved both the insertion of the chest drain and the completion of the intervention. If the participant expressed their desire to discontinue the intervention, this was also recorded as the endpoint of the scenario.
Team performance | Through study completion, an average of 8 minutes per scenario
  The OTAS tool (Observational Teamwork Assessment for Surgery) is a validated scale that is commonly used to assess team performance in surgery. It is a structured observation tool that allows for the assessment of teamwork in the operating room setting, and it has been shown to have good inter-rater reliability and construct validity.
  The tool can also be used to compare the performance of individual team members and to determine how the use of technology influences cognitive load and individual perspective performance. For example, studies have used the OTAS tool to evaluate the impact of laparoscopic surgery on team performance and to determine how the use of surgical robots affects teamwork and communication in the operating room.
Team performance | Through study completion, an average of 8 minutes per scenario
  The T-SAW-C Tool (Teamwork Skills Assessment for Ward Care) was used by observers to assess teamwork during the simulated scenarios. This tool measures various aspects of teamwork, such as communication, coordination, and cooperation, and has been validated for use in healthcare settings. By including this information, it clarifies the measurement tool being used to assess the specific outcome measure of interest.
Team workload | Through study completion, an average of 8 minutes per scenario
  The NASA Task Load Index (TLX) is a subjective multidimensional assessment tool that rates perceived workload in order to assess a task, system, or team's effectiveness or other aspects of performance. It uses a Likert scale with six domains, each attributed a weight ranging from 0 to 5. The scale ratings are scored based on where the user marked the scale. Tick marks range from 0 to 100 by 5 point increments, and scores are given for the tick at or immediately above the mark. Higher scores indicate a greater perceived workload.

CONTACTS AND LOCATIONS:
Overall Officials: James Kinross, PhD FRCS, Principal Investigator — Senior Lecturer in Surgery and Consultant Surgeon
Locations (1):
- Department of Surgery and Cancer Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Lawson J, Martin G, Guha P, Gold M, Nimer A, Syed S, Kinross J. Effect of Mixed Reality on Delivery of Emergency Medical Care in a Simulated Environment: A Pilot Randomized Crossover Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2330338. doi: 10.1001/jamanetworkopen.2023.30338. PMID 37639272